CLINICAL TRIAL: NCT00281255
Title: Allopurinol and Cardiac Function Pilot Study in Idiopathic Dilated Cardiomyopathy
Brief Title: Intravenous Allopurinol to Improve Heart Function in Individuals With Dilated Cardiomyopathy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Infeasible
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Thomas Cappola, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 353; K23HL071562 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Diseases; Cardiomyopathy, Dilated; Heart Diseases; Heart Failure, Congestive
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathy, Dilated; Heart Diseases; Heart Failure | interventions — Allopurinol; Dobutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- allopurinol (Experimental)
  Interventions: Drug: Allopurinol; Drug: Dobutamine
- placebo (Placebo Comparator)
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Allopurinol
  Arms: allopurinol
Drug: Dobutamine

SUMMARY:
This study will determine whether an acute infusion of intravenous allopurinol improves the inotropic response to dobutamine in patients with idiopathic dilated cardiomyopathy (DCM) as measured by cardiac magnetic resonance imaging (CMR).

DETAILED DESCRIPTION:
BACKGROUND:

DCM is a poorly understood cause of systolic heart failure and is the most common indication for heart transplantation in the United States. Despite advances in medical and device therapy, the 5-year mortality of patients with DCM remains near 50%.

Oxidative stress, an imbalance between the formation and degradation of free radicals within the myocardium, contributes to metabolic derangements in patients with DCM. The enzyme xanthine oxidase (XO), a potent source of oxidative stress, is expressed in the failing heart, and it uncouples cardiac energy consumption from cardiac contraction in the setting of chronic heart failure. These effects can be reversed by inhibiting XO with the XO inhibitor allopurinol, resulting in a marked increase in cardiac efficiency. These findings provide a rationale for using allopurinol to enhance cardiac function in DCM. However, there is little data on the effects of allopurinol therapy on cardiac function. Therefore, the primary aim of this study is to determine whether an acute infusion of intravenous allopurinol improves the inotropic response to beta-adrenergic stimulation in patients with idiopathic DCM.

Decreased beta-adrenergic responsiveness is a characteristic feature of DCM that is attributable in part to decreased expression of the beta 1-receptor in chronic heart failure, as well as dysregulation of down-stream signaling pathways. Improvement in beta-adrenergic responsiveness is a useful surrogate marker for long-term improvement in cardiac structure, function, and decreased cardiac events. Traditionally, invasive hemodynamic monitoring using pressure and pressure/volume catheters has been the method of choice to quantify the inotropic response in heart failure. However, newly developed magnetic resonance imaging (MRI) techniques now allow precise assessment of the inotropic response non-invasively. Studies have shown that tagged CMR is a reproducible, noninvasive method to quantify the inotropic response to the beta 1 agonist dobutamine in individuals with structurally normal hearts. Specifically, radial strain (E1) and circumferential strain (E2) are measured at increasing doses of dobutamine using tagged CMR. Changes in these strain parameters, now referred to as delta E1 and delta E2, are precise measurements of the beta-inotropic response.

DESIGN NARRATIVE:

An estimated 20 patients with DCM will be randomized in a 1:1 ratio fashion to receive allopurinol or placebo. The primary aim of this investigation is to determine whether an acute infusion of intravenous allopurinol improves the inotropic response to dobutamine in patients with idiopathic DCM as measured by CMR. Specifically, the study will test the hypothesis that a single dose of intravenous allopurinol, compared to placebo, enhances delta E1 and delta E2. Secondary aims of this study are as follows: 1) to determine whether the response to allopurinol is associated with baseline XO activity and levels of natriuretic peptides (investigators predict that augmentation in delta E1 and delta E2 will correlate positively with baseline plasma uric acid and plasma B-type natriuretic peptide [BNP]); and 2) to demonstrate that tagged dobutamine CMR is a useful non-invasive technique to assess pharmacologic responses in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic cardiomyopathy (defined by an ejection fraction less than or equal to 35% that has been assessed by any method within 6 months prior to study entry AND no evidence of coronary artery disease, as determined by coronary angiography or stress perfusion imaging within 2 years prior to study entry)
* New York Heart Association (NYHA) Class I - II heart failure
* Stable heart failure medication for at least 1 month prior to study entry
* Able to lie flat for 45 minutes

Exclusion Criteria:

* History of poorly controlled hypertension and concentric left ventricular hypertrophy on echocardiography suggesting hypertensive cardiomyopathy
* History of biopsy-proven myocarditis
* Peripartum cardiomyopathy
* Allopurinol therapy within the 6 months prior to study entry
* Allopurinol allergy
* Contraindication to allopurinol because of concomitant therapy with one of the following: azathioprine, cyclophosphamide, dicumarol, uricosuric agents (e.g., probenecid), ampicillin, amoxicillin, chlorpropamide, or cyclosporine
* Acute gout
* Estimated creatinine clearance less than 20 ml/min
* Total bilirubin greater than 2 times upper limit of normal
* Serum aspartate AST or alanine ALT greater than 3 times the upper limit of normal
* White blood cell count less than 2,000
* Platelet count less than 80,000
* Hemoglobin less than 8 mg/dl
* Use of intravenous inotropes
* History of untreated symptomatic ventricular tachycardia
* History of sustained ventricular tachycardia induced by dobutamine
* Contraindication to MRI because of one of the following:

  1. Starr-Edwards pre-6000 series prosthetic valves or prosthetic valves for which model can not be determined
  2. Implanted pacemaker
  3. Implanted cardioverter-defibrillator intracranial aneurysm clips
  4. Other implanted medical devices that are known to be MRI incompatible (e.g., cochlear implants and spinal stimulators)
  5. History of foundry-work that could create ocular metallic fragments
* Hospitalization at least 1 month prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
radial and circumferential strain after infusion of allopurinol as measured by cardiac MRI (measured at Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Cappola, Study Chair — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States